CLINICAL TRIAL: NCT03789903
Title: Amniotic Fluid Lactate in Predicting Latency in Perterm Premature Rupture of Membranes
Brief Title: Amniotic Fluid Lactate in Perterm Premature Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, Principal Investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ain shams maternity hos
Record Dates: First submitted 2018-12-26; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Rupture of Membranes; Premature
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: amniotic fluid lactate — AF lactate

SUMMARY:
AF lactate level could help in predicting the duration from ROM till delivery

ELIGIBILITY:
Inclusion Criteria:

1. women with PPROM
2. GA between 24 to 34 weeks

Exclusion Criteria:

1. chorioamnionitis
2. previous Preterm labor
3. abruptio placentae
4. UTI ,pyelonephritis

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
latency period | upto 48 hours
  duration from ROM till the occurrence of active labor

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt